CLINICAL TRIAL: NCT03026699
Title: Refining and Testing the Electronic Social Network Assessment Program (eSNAP)
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Utah (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: MCC-18378; R03CA201684-01 (NIH)
Record Dates: First submitted 2017-01-12; First posted 2017-01-20 (Estimated); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Brain Cancer
Keywords: Brain; Nervous system; Neuro-oncology; Caregivers; Cancer patient; Family caregivers; Brain tumors; Quality of life; Stress; Social support; Feasibility; Electronic Social Network Assessment Program (eSNAP)
MeSH Terms: conditions — Brain Neoplasms; Neurologic Manifestations | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Intervention - Primary Brain Tumor: eSNAP Intervention Plus Questionnaires: Family caregivers of primary brain tumor patients.
  Interventions: Behavioral: eSNAP; Behavioral: Questionnaires
- Intervention - Secondary Brain Tumor: eSNAP Intervention Plus Questionnaires: Family caregivers of secondary brain tumor patients.
  Interventions: Behavioral: eSNAP; Behavioral: Questionnaires
- Control - Primary Brain Tumor: Questionnaires Only Control: Family caregivers of primary brain tumor patients.
  Interventions: Behavioral: Questionnaires
- Control - Secondary Brain Tumor: Questionnaires Only Control: Family caregivers of secondary brain tumor patients.
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: eSNAP — Participants in the intervention group will then be given a tablet loaded with the eSNAP application and asked to create a visualization of their social networks. Upon completion, participants will be asked to review their ecomaps and complete the user experience questionnaire.
  Other Names: Electronic Social Network Assessment Program
  Groups: Intervention - Primary Brain Tumor; Intervention - Secondary Brain Tumor
Behavioral: Questionnaires — Participants will complete demographics and baseline (T1; baseline) questionnaires. For all participants Time 2 (T2; 3 week) and Time 3 (T3; 6 week) questionnaires will be completed either by phone, mail, or email (depending on participant preference) to assess longer-term effects of eSNAP on outcomes versus controls.

SUMMARY:
The purpose of the study is to learn more about neuro-oncology caregivers' quality of life and how friends and families help neuro-oncology cancer caregivers at different times during treatment.

DETAILED DESCRIPTION:
Former Aim 1: Refine eSNAP data-gathering and visualization prototypes based on evaluations of user experience, including usability, satisfaction and applicability. The refining process was completed at the University of Utah.

Aim 2: Test the feasibility of implementing eSNAP in a neuro-oncology clinical setting and collect preliminary effectiveness data of eSNAP on Family Caregiver outcomes, including quality of life and stress, and mediators (Family Caregiver social support utilization and burden). The feasibility process will take place at Moffitt Cancer Center.

This study will be a 2x2 longitudinal design. Caregivers of primary brain tumor patients will be compared to caregivers of patients with secondary brain tumors (brain metastases) to determine if there is something unique about the cancer-specific duties of primary versus secondary brain tumors that could impact the effectiveness of the eSNAP application. An intervention group will be compared to a control group for both types of caregivers. Participants will be randomized 2:1 for the intervention and control. All caregivers will be followed for 6 weeks and will be asked to complete questionnaires at 3 time points; caregivers in the intervention group will also be asked to use the eSNAP application at time 1, which will be available to them for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Family caregiver of a patient with primary or secondary brain tumor
* Age 18 years or older
* Able to speak and write English

Exclusion Criteria:

* Does not meet the Inclusion Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be family caregivers recruited from the Moffitt Cancer Center Radiation Oncology Clinic.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Questionnaire Participation Among Participant Groups | 6 weeks per participant
  Feasibility 1: Recruitment rates per group.
Retention of Participants Among Participant Groups | 6 weeks per participant
  Feasibility 2: Retention rates per group.

SECONDARY OUTCOMES:
Stress and Coping - Quality of Life Among Participant Groups | 6 weeks per participant
  Although not reaching adequate power to detect differences, planned analysis will allow investigators to estimate effect size of eSNAP at baseline as well as the effect of cancer type. (Power analysis conducted in G*Power for ANOVA using effect size 0.2 a=.05 for 3 groups for power of 0.80 requires a sample of 246.) ANOVA will be conducted to determine if groups vary on stress and quality of life at baseline. Growth-curve analysis will be used to identify potential preliminary differences in the eSNAP group over time.
Perceived Social Support - Quality of Life Among Participant Groups | 6 weeks per participant
  Chi square and generalized linear model (GLM) will be used to analyze utilization of support services differences.
Incidence of Clinic Disruption | 6 weeks per participant
  Incidence of clinic disruption per participant group.
Incidence of Problems with eSNAP implementation | 6 weeks per participant
  Chi square and generalized linear model (GLM) will be used to analyze trends in satisfaction or time spent on ecomapping/eSNAP.

CONTACTS AND LOCATIONS:
Overall Officials: Maija Reblin, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Reblin M, Ketcher D, Forsyth P, Mendivil E, Kane L, Pok J, Meyer M, Wu YP, Agutter J. Feasibility of implementing an electronic social support and resource visualization tool for caregivers in a neuro-oncology clinic. Support Care Cancer. 2018 Dec;26(12):4199-4206. doi: 10.1007/s00520-018-4293-z. Epub 2018 Jun 12. PMID 29948397
- See also: Moffitt Cancer Center Clinical Trials website — https://moffitt.org/clinical-trials-research/